CLINICAL TRIAL: NCT04056416
Title: Physical Activity Promotion in Children and Adolescents With Single Ventricle Physiology (MedBike)
Acronym: MedBike
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00057730
Record Dates: First submitted 2019-04-25; First posted 2019-08-14 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Congenital Heart Defect; Hypoplastic Left Heart Syndrome; Physical Activity
MeSH Terms: conditions — Heart Defects, Congenital; Hypoplastic Left Heart Syndrome; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HIIT Exercise Program (Experimental): Exercise on a MedBIKE 3 times a week for 8 weeks with pre- and post-CPET testing, questionnaires and qualitative interviews.
  Interventions: Device: MedBIKE

INTERVENTIONS:
Device: MedBIKE — A MedBIKE will be installed into a participants home and connected to clinicians via telehealth for monitoring during exercise sessions. Sessions will be based on standardized guidelines for aerobic exercise. Heart rate, ECG, oxygen saturation and rating of perceived exertion will be monitored throughout the session.

SUMMARY:
Single ventricular (SV) heart was a uniformly fatal condition before the advances in surgical treatment in 1980. In the present era, 5-year survival rate with SV is 75%, with some centers, including the Stollery Children's Hospital reporting higher survival. Although mortality remains a major concern, the research focus has shifted to management of late complications as well as improving patient physical and mental health related quality of life issues. Children with SV have reduced exercise tolerance and this is progressive through adulthood. Recent advances in remote health assessment and telehealth systems have allowed the development of medically supervised home graduated physical training for adult cardiac patient rehabilitation. To our knowledge, the application of these technologies has not been applied to SV patients. The long term goal is to use this technology to improve patient exercise capacity and to positively influence parental and patient perceptions of the patient's physical ability.

DETAILED DESCRIPTION:
Children with single ventricular (SV) heart were a uniformly fatal condition prior to descriptions of surgical palliation in 1980 that results in a Fontan circulation with single ventricle physiology. In the present era, 5-year survival is 75% in multicenter studies, with some centers including the Stollery Children's Hospital reporting higher survival. Although mortality remains a challenge for this population, the research focus has shifted towards optimizing management of late complications as well as improving patient physical and mental health-related quality of life issues. Children with SV have decreased exercise tolerance and the reduction is progressive through adolescence and into adulthood. Physical factors contributing to decreased exercise tolerance in the Fontan patient include cardiovascular inefficiencies and the loss of peripheral lean muscle mass and efficiency from deconditioning. Recently, Cordina et al. has shown that an intensive exercise regiment can improve muscle strength and mass, cardiac output and exercise capacity in adults with Fontan circulation. The majority of published outcomes from exercise training in patients with congenital heart disease (CHD) have resulted in increased measured exercise capacity with no apparent negative effect. Although the link between improved exercise capacity and improved patient quality of life remains controversial, participation in an aerobic exercise regimen leads to improved health-related quality of life.

Aside from physical limitations to their exercise capacity, Fontan patient self-confidence toward physical activity is low, as is exercise participation. Studies indicate that amongst youth with CHD, low self-confidence may be a more important predictor of participation than the severity of the disease. Parental overprotection is a common finding in children with CHD with a lasting impact on patient self-confidence and anxieties toward physical activity well into adulthood. Alteration of patient and parental perception and anxieties toward participation in physical activity may improve compliance to exercise training and encourage more positive patient perceptions toward healthy lifestyle habits, including frequent physical activity participation.

Recent technological advances in remote health assessment capabilities and telehealth systems have allowed the development of medically supervised home graduated physical training for adult cardiac patient rehabilitation. The application of such technologies to pediatric congenital heart patients has not been tested. In collaboration with Prof. Boulanger at the Advanced Man Machine Interface Laboratory at the University of Alberta, a custom pediatric remote bike ergometer (MedBike) was developed. This technology provides the medical supervisor with a live-feed of patient video/audio, electrocardiograph (ECG), blood pressure (BP) and blood oximetry signals while enabling remote determination of patient work load through the bike ergometer. The long-term goal is to use this technology to improve patient exercise capacity and to positively influence patient and parental perceptions of the patient's physical ability.

Stage 2 (HIIT exercise program): The investigators will evaluate the safety and efficacy of an 8-week, 3 times per week supervised HIIT exercise program in patients with SV physiology.

All eligible patients will undergo a full cardio pulmonary exercise testing (CPET) and anthropometry assessment of lean muscle mass prior to exercise training and at the end of the training period. Understanding that a patient's CPET results may change over time, subjects who participated in Stage 1 of the study will be invited back to undergo a new baseline CPET to ensure the reliability of the data.

A MedBike will be installed in the participant's home. Members of the MedBike team at the University of Alberta will be responsible for installation, set-up, and training with regards to participant use of the MedBike. Installation, set-up, and training will occur at a time that is convenient for the participant and their caregivers. The patients will exercise in the convenience of their home with tele-health link that includes a live video and audio feed to the supervisor workstation at the University of Alberta. The HIIT program described above will be applied. The supervisor will have the ability to modify the program intensity during each session based on the perceived difficulty or ease of it and the results of the baseline CPET. The exercise sessions in their home will be also be supervised in-person by the patient's caregiver. Given that no adverse events or safety concerns arose in Stage 1B of the study, the patient will be supervised remotely by a member of the MedBike team capable of reading ECG data. The investigators will document any adverse effects from the 240 training sessions during the study.

Exercise sessions will be based on standardized guidelines for aerobic exercise (ACSM's guidelines for exercise testing and prescription 2013). Heart rate, ECG, oxygen saturation and rating of perceived exertion will be monitored during each session.

Any adverse events such as profound desaturation (oxygen saturations fall of > 10% points for greater than 1 min, chest pain and ECG changes consistent with ischemia (ST depression or elevation in 2 consecutive leads), development of tachyarrhythmia (atrial or ventricular) and any bike injury, will result in immediate stoppage of exercise regimen and evaluation by the remote supervisor with access to medical personnel..

The impact of the exercise program on patient and parental perceptions of the patient's physical capacity will be evaluated using qualitative methods, as well as health related quality of life questionnaires. Patient and parents will be interviewed prior to, and at the end of, the exercise training as to their perceptions of the influence of physical activity in the presence of complex CHD.

ELIGIBILITY:
Inclusion Criteria:

* single ventricle patients with Fontan circulation

Exclusion Criteria:

* Cardiac arrhythmias
* Persistent low resting oxygen saturation of < 85%
* Severe ventricular dysfunction on most recent clinical echocardiogram
* Patients with reports of chest pain on exertion
* Restricted exercise by cardiologist

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2020-03-19 (Actual); Study Completion 2022-11-09 (Actual)

PRIMARY OUTCOMES:
Exercise capacity | Pre- VO2 max performed 1 week before 24 HIIT exercise sessions and within 1 week after last session
  Exercise capacity assessed as the change in max VO2 pre- vs. post- completion of the HIIT exercise program. Hypothesis- we will observe an increased in VO2 max of 15%.

SECONDARY OUTCOMES:
Qualitative interviews to determine the perception of exercise in CHD patient | Pre-interview conducted within 2 weeks of beginning 24 HIIT exercise sessions and post interview conducted within 2 weeks after last session
  Patient and parental perception of a CHD patient's safety and limitations while performing physical activity through a successful physical rehabilitation program
Number of participants with exercise program specific adverse events | Data on acute events are recorded only during the study regiment (24 HIIT sessions); 8 weeks total
  Adverse events to determine the safety profile of the exercise program

CONTACTS AND LOCATIONS:
Overall Officials: Nee Khoo, MD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-02-24): https://cdn.clinicaltrials.gov/large-docs/16/NCT04056416/Prot_SAP_ICF_000.pdf